CLINICAL TRIAL: NCT06637761
Title: Clinical and Radio-graphic Evaluation of Bio-active Bio-ceramic (Neo MTA 2) Versus White MTA Used as Coronal Plug Material in Revascularization of Non-vital Immature Permanent Anterior Teeth: A Randomized Clinical Trial
Brief Title: Clinical and Radio-graphic Evaluation of Non-staining Bio-active Bio-ceramic (Neo MTA 2) in Revascularization
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ola mourad, Assisstant lecturer in pediatric dentistry department, faculty of dentistry, Misr University for sience and technology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cairo U Clinical
Record Dates: First submitted 2024-09-19; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mineral Trioxide Aggregate
Keywords: bioactive bioceramic; discoloration; revascularization; mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple(Patients, radio-graphic outcome assessor(s), and statisticians) will be blinded in this study.
  Blinding to participant: will not know either the intervention or the comparative will be applied to their teeth Blinding to outcome assessor: to overcome detection bias Blinding to statisticians: to overcome bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (Experimental): NeoMTA 2
  Manipulation and mixing will be done according to manufacturer instructions:
  * 1 scoop (0.1gm) of NeoMTA 2 Powder will be dispensed on a glass slab. Then two drops of NeoMTA 2 Gel will be dispensed next to the powder.
  * Gradually as much Gel as necessary will be added to the Powder to achieve the desired consistency. The Gel will be incorporated by spatula-ting the Powder/Gel mixture firmly against the glass slab to ensure all of the Powder is thoroughly witted by the Gel.
  Interventions: Drug: NeoMTA2
- Group II (Active Comparator): White mineral trioxide aggregate
  * One spoon of powder and one drop of distilled water are dispensed on a sterile glass slab.
  * A metal spatula will be used to gradually mix the liquid and powder together for 30 seconds to ensure full wetting of the powder particles and to obtain a consistency similar to wet sand.
  * 3-4 mm of white MTA will be placed over the clot carefully by using an amalgam carrier.
  The mix will be placed over the collagen matrix 2mm beneath the clinical cement-enamel junction.
  Interventions: Drug: WMTA

INTERVENTIONS:
Drug: NeoMTA2 — Bio-active bio-ceramic mineral trioxide aggregate
  Other Names: Nu smile,USA
  Arms: Group I
Drug: WMTA — White Mineral trioxide aggregates
  Other Names: Angulus, Brazil
  Arms: Group II

SUMMARY:
The study will compare the clinical and radio-graphic performance of newly introduced non-staining bio-active bio-ceramic (Neo MTA 2) versus White MTA used as coronal plug material in revascularization of non-vital immature permanent anterior teeth.Visual examination, palpation, A measuring scale in digital radio-graph software (DIGORA for Windows software) will be used for evaluation.

DETAILED DESCRIPTION:
Mineral trioxide aggregate (MTA) has been widely used in revascularization procedures for coronal sealing in more than 85% of studies for privilege of bio compatibility, good sealing properties, and marginal adaptation. However, its poor handling characteristics and potential coronal discoloration effects are the major disadvantages of using mineral trioxide aggregate.

Although white MTA (WMTA) has been developed to overcome the tooth discoloration caused by the application of grey MTA, several in vivo and in vitro studies have also reported tooth discoloration after using WMTA.

To overcome the problems associated with WMTA, a new modification was introduced to the market called NeoMTA 2 as a new hope to overcome the discoloration problem. NeoMTA 2 provides easier handling, shorter setting time, and better color. The lack of post-operative discoloration problems was mainly due to the absence of Bismuth oxide in NeoMTA.

up to date, no clinical trials have reported the clinical and radio-graphic outcomes after revascularization of non-vital immature permanent anterior teeth using Neo MTA 2. Thus, the present study aims to evaluate and compare clinically and radio-graphically the effect of using two different coronal plug materials (Neo MTA 2 versus White mineral trioxide aggregate) in revascularization of non-vital immature permanent anterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative patient/ compliant parents or guardians
* Patients free from any systemic diseases that hinder the normal healing process according to parental history
* Necrotic immature permanent anterior teeth
* Enough coronal portion of teeth that does not necessitate post and core for final restoration

Exclusion Criteria:

* Patients having an allergy to medicament and antibiotics necessary to complete the procedure
* Teeth with internal or external root resorption
* Uncooperative patients/ in-compliant parents or guardians
* Laxative injuries
* Avulsed tooth after re-plantation
* Compromised remaining coronal structure

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2024-10-05 (Estimated); Primary Completion 2025-10-06 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Discoloration | 1 year
  Using shade guide (VITA classical)

OTHER OUTCOMES:
swelling | 1 year
  Clinical examination (Visual examination and palpation of the labial vestibule and the palatal area related to every affected tooth)

CONTACTS AND LOCATIONS:
Overall Officials: Youssef, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No